CLINICAL TRIAL: NCT02524418
Title: Prospective Evaluation of the Clinical Utility of Endoscopic Retrograde Cholangiopancreatography (ERCP) Guided Cholangiopancreatoscopy With the SpyGlass DS.
Brief Title: Clinical Utility of ERCP Guided Cholangiopancreatoscopy With the SpyGlass DS
Acronym: SPYDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 483-2006
Record Dates: First submitted 2015-08-07; First posted 2015-08-14 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Biliary Tract Disease
Keywords: Main Pancreatic Duct
MeSH Terms: conditions — Biliary Tract Diseases | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cholangiopancreatoscopy (Other): A standard of care Endoscopic Retrograde Cholangiopancreatoscopy (ERCP) will be performed using the Spyglass DS. The clinical outcomes will be collected and analyzed.
  Interventions: Procedure: Cholangiopancreatoscopy

INTERVENTIONS:
Procedure: Cholangiopancreatoscopy — An ERCP with cholangioscopy/pancreatoscopy will be performed using the Spyglass DS. Clinical outcomes will be collected and analyzed.
  Other Names: ERCP

SUMMARY:
This is a prospective evaluation of the clinical utility of the new cholangioscopy platform SpyGlass DS. The aims of this study are to prospectively document the clinical utility and technical aspects of ERCP with cholangioscopy and/or pancreatoscopy in the diagnosis and management of pancreatic-biliary disorders.

DETAILED DESCRIPTION:
Cholangioscopy allows for direct visualization of the bile and pancreatic duct. In 2006, the SpyGlass Direct Visualization System for per-oral cholangiopancreatoscopy was introduced and since then has been shown to provide incremental diagnostic and therapeutic benefits. The main limitations of the original SpyGlass platform are fiber optic visualization system, limited tip angulation, square cut Spy scope tip, and complex multi-component setup. A new generation cholangioscopy platform, SpyGlass DS is currently in clinical use. The new system addresses many of the shortcomings of old platform including digital optics, improved tip angulation, tapered tip and simplified set up. It is unclear at this time whether this technical improvement will translate into better outcomes. Therefore, the investigators want to study the clinical utility of SpyGlass DS by prospectively collecting data on the clinical outcomes of patients undergoing cholangioscopy with Spyglass DS as part of their routine medical care.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have been scheduled to undergo a cholangiopancreatoscopy as routine clinical care

Exclusion Criteria:

* failure to provide informed consent
* any contraindications to endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter V Draganov, MD, Principal Investigator — University of Florida
Locations (1):
- Shands at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cholangiopancreatoscopy
Started | 88
Completed | 75
Not Completed | 13

BASELINE CHARACTERISTICS:
Population: 88 subjects signed consent but in 13 subjects a Spyglass examination was not done because of the lack of indication after performing standard cholangiography or pancreatography
Arm/Group | Cholangiopancreatoscopy
Number analyzed (Participants) | 75
Age, Continuous [Mean (Full Range); unit: years] | 66 [22 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedure Technical Success
Description: The performance of the Spyglass DS during the endoscopy will be based on the ability to reach the target site, obtain samples, and to deliver therapeutic intervention.
Time Frame: Day 1
Population: Five of the subjects had both Cholangioscopy and Pancreatoscopy. The results of these procedures were recorded and analyzed separately
Measure: Number; unit: participants
Groups:
- Cholangioscopy: A standard of care Endoscopic Retrograde Cholangiopancreatoscopy (ERCP) will be performed using the Spyglass DS. The clinical outcomes will be collected and analyzed.
  Cholangiopancreatoscopy: An ERCP with cholangioscopy/pancreatoscopy will be performed using the Spyglass DS. Clinical outcomes will be collected and analyzed.
- Pancreatoscopy: These are the subjects who had evaluation of their pancreas ducts during the Spyglass ERCP
Arm/Group | Cholangioscopy | Pancreatoscopy
Number analyzed (Participants) | 75 | 5
participants | 70 | 3

2. Secondary Outcome: Time to Set-up the Spyglass DS for the Procedure
Description: The time it takes to set up the Spyglass DS and related equipment for the procedure.
Time Frame: approximately 2 hours
Population: In 20 procedures, the Spyglass equipment set up was done after ERCP started and this time was recorded. The Investigators did not record the set up time for the other procedures.
Measure: Mean (Full Range); unit: minutes
Arm/Group | Cholangiopancreatoscopy
Number analyzed (Participants) | 20
minutes | 5 [2.61 to 7.39]

3. Secondary Outcome: Measurement of Total Procedure Time Using the Spyglass DS
Description: Time in minutes will be calculated for completing the procedure with the Spyglass DS.
Time Frame: approximately 2 hours
Population: 83 Spyglass procedures were conducted on the 75 participants
Measure: Mean (Full Range); unit: minutes
Units Other Than Participants: number of Spyglass procedures
Arm/Group | Cholangiopancreatoscopy
Number analyzed (Participants) | 75
Number analyzed (number of Spyglass procedures) | 83
minutes | 64.3 [39.1 to 89.4]

4. Secondary Outcome: Measurement in Minutes for Spyglass DS Diagnostic Maneuvers
Description: The time it takes to perform the diagnostic maneuvers with the SpyGlass DS measured in minutes.
Time Frame: approximately 2 hours
Population: 83 Spyglass procedures were performed on the 75 participants
Measure: Mean (Full Range); unit: minutes
Units Other Than Participants: number of Spyglass Proceudres
Arm/Group | Cholangiopancreatoscopy
Number analyzed (Participants) | 75
Number analyzed (number of Spyglass Proceudres) | 83
minutes | 27.5 [10.8 to 44.2]

5. Secondary Outcome: Measurement in Minutes for Spyglass DS Therapeutic Maneuvers
Description: The time it takes to perform the therapeutic maneuvers with the SpyGlass DS in cases sampling was attempted measured in minutes.
Time Frame: approximately 2 hours
Population: For the 75 participants in the study, 83 procedures were completed. Of the 83 procedures, sampling was attempted on 37 procedures in 27 participants.
Measure: Mean (Full Range); unit: minutes
Units Other Than Participants: Number of Procedures analyzed
Arm/Group | Cholangiopancreatoscopy
Number analyzed (Participants) | 27
Number analyzed (Number of Procedures analyzed) | 37
minutes | 12.1 [5.76 to 18.44]

6. Secondary Outcome: Number of Cholangioscopic Exams That Detected Ductal Stones
Description: The abnormalities found during the procedure, such as ductal stones.
Time Frame: Day 1
Population: There were a total of 78 Cholangioscopic examinations in the 70 subjects in this study; 35 exam found stones. Where as in the Pancreatoscopy arm 5 participants were evaluated with only 3 exams being evaluable..
Measure: Number; unit: exams
Units Other Than Participants: total number of exams
Groups:
- Pancreatoscopy: Subject who had a Pancreatoscopy as part of their ERCP
Arm/Group | Cholangioscopy | Pancreatoscopy
Number analyzed (Participants) | 70 | 5
Number analyzed (total number of exams) | 78 | 3
exams | 35 | 2

7. Secondary Outcome: Strictures Found During the Procedure Will be Measured
Description: The abnormalities found during the procedure, such as strictures.
Time Frame: Day 1
Population: A total of 78 Cholangioscopic examinations were attempted
Measure: Number; unit: strictures found
Units Other Than Participants: attempted Cholangioscopic exams
Arm/Group | Cholangioscopy
Number analyzed (Participants) | 75
Number analyzed (attempted Cholangioscopic exams) | 78
strictures found | 27

8. Secondary Outcome: Spybite Sampling Attempts Per Procedure
Description: The mean number of attempts per procedure
Time Frame: Day 1
Population: Of the 70 Cholangioscopy participants in the study only 44 participants had non-stone lithotripsy-related indications. Spyglass sampling was attempted in 36 procedures.
Measure: Mean (Full Range); unit: sampling attempts per procedure
Units Other Than Participants: Number of procedures analyzed
Arm/Group | Cholangioscopy
Number analyzed (Participants) | 44
Number analyzed (Number of procedures analyzed) | 36
sampling attempts per procedure | 3.94 [2.47 to 5.41]

9. Secondary Outcome: Number of Participants With Successful Removal of the Biliary or Pancreas Stones
Description: The successful removal of the biliary or pancreas stones will be determined by the need for additional procedures.
Time Frame: Day 1
Population: Spyglass-guided stone therapy was attempted in 26 patients with biliary stones
Measure: Number; unit: participants
Arm/Group | Cholangioscopy
Number analyzed (Participants) | 26
participants | 24

ADVERSE EVENTS:
Arm/Group | Cholangiopancreatoscopy
Serious Adverse Events (participants affected / at risk) | 1/75
Other Adverse Events (participants affected / at risk) | 3/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholangiopancreatoscopy (N=75)
periampullary perforation (Gastrointestinal disorders) | 1 (1) — Serious AE with periampullary perforation caused by biliary sphincterotomy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholangiopancreatoscopy (N=75)
mild Post ERCP pancreatitis (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No